CLINICAL TRIAL: NCT05837689
Title: Minimal Residual Disease Quantification by Next-generation Sequencing in Pediatric B-ALL Children Patients Treated With Blinatumomab Consolidation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiaojun Xu (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Xu, Principal investigator, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Other Study IDs: 2023-IRB-0062-P-01
Record Dates: First submitted 2023-03-31; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Blinatumomab — IV

SUMMARY:
A retrospective analysis to investigate pediatric B-cell acute lymphoblastic leukemia patients who were treated with blinatumomab for consolidation, and who were detected as minimal residual disease (MRD) positive by next generation sequencing (NGS). The efficacy of blinatumomab clearing MRD detected by NGS will be analyzed, in order to see the potential of using NGS to guide MRD eradication by blinatumomab.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with B cell precursor acute lymphoblastic leukemia
* Patients who received blinatumomab for consolidation
* Patients who were detected MRD positive by NGS before initiation of blinatumomab treatment

Exclusion Criteria:

* Patients without data of NGS detection after receiving blinatumomab treatment

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric BCP-ALL patients who were treated in our institution since Oct 2021
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
MRD clearance rate (MRD<0.00001%) | before blinatumomab initiation (baseline), Day 15 of blinatumomab treatment, Day 29 of blinatumomab treatment
  The change of MRD will be detected by NGS, with sensitivity of 0.00001% and 0.01%, respectively